CLINICAL TRIAL: NCT03426280
Title: Activity Therapy After Kidney Transplant: A Pilot Study
Brief Title: Activity Therapy After Kidney Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to Covid-19 health emergency
Sponsor: Stanford University (Other)
Collaborators: Apple Inc. (Industry)
Responsible Party: Principal Investigator, Xingxing Shelley Cheng, Clinical Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44663
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Kidney Transplant; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple Watch (Experimental): Clinic pharmacists will issue Apple Watches to study arm patients and teach them the usage of the Activity app. In addition to usual care, these patients will each receive an in-person 3-minute coaching session during clinic visit at 2, 4, 6 and 12 months.
  Interventions: Device: Apple Watch Series 1
- Usual Care (No Intervention): Usual care.

INTERVENTIONS:
Device: Apple Watch Series 1 — Clinic pharmacists will issue Apple Watches to study arm patients and teach them the usage of the Activity app. In addition to usual care, these patients will each receive an in-person 3-minute coaching session during clinic visit at 2, 4, 6 and 12 months.
  Arms: Apple Watch

SUMMARY:
To combat post-transplant weight gain, we seek to expand Stanford Kidney Transplant's multidisciplinary platform to include physical activity monitoring and coaching using the Apple Watch.

ELIGIBILITY:
Inclusion Criteria:

* All adults (18 years) who undergo kidney transplant at Stanford.

Exclusion Criteria:

* Poor vision with inability to use Apple Watch
* Permanently unable to ambulate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Activity Level (daily caloric consumption) | 1 year
% Days using Apple Watch | 1st year of transplant

SECONDARY OUTCOMES:
Weight | 1st year of transplant
Hemoglobin A1c | 1st year of transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinic, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No